CLINICAL TRIAL: NCT06386289
Title: Safety, Performance and Lesion Evaluation of Neurothrombectomy Using CEREGLIDE 92 Intermediate Catheter: A Prospective Multi-Center Single-Arm IDE Trial (SPLENDID)
Brief Title: Safety, Performance of CEREGLIDE 92 Intermediate Catheter in Treatment of Acute Ischemic Stroke
Acronym: SPLENDID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a change in innovation strategy
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNV202202; CNV202202 (Other: Cerenovus, Part of DePuy Synthes Products, Inc.)
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): Mechanical Thrombectomy
  Interventions: Device: Cereglide 92

INTERVENTIONS:
Device: Cereglide 92 — Aspiration of cerebral large vessels occlusions

SUMMARY:
The device is indicated for use in the revascularization of patients with acute ischemic stroke secondary to intracranial large vessel occlusive disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute ischemic stroke.
* NIHSS ≥6
* Baseline mRS ≤ 2
* Completed informed consent.

Exclusion Criteria:

* Known pregnancy.
* Life expectancy less than 90 days prior to stroke onset.
* Known Diagnosis of Dementia
* Treatment with heparin within 48 hours.
* Clinical history, past imaging or clinical judgement suggest that the intracranial occlusion is chronic.
* Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
* Baseline CT or MRI showing mass effect
* Concurrent sino-venous thrombosis
* Currently participating in an investigational (drug, device, etc.) clinical trial, excluding trials in observational, natural history, and/or epidemiological studies not involving intervention and that will not confound study endpoints. Sponsor approval is required.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
First pass reperfusion | Intraprocedural
  First pass reperfusion (eTICI ≥ 2b50 without additional therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Froehler, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Brian Jankowitz, MD, Principal Investigator — JFK University Medical Center; Ansaar Rai, MD, Principal Investigator — West Virginia University

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA)
Access Criteria: Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu